CLINICAL TRIAL: NCT00537901
Title: First-Line Bevacizumab and Chemotherapy in Metastatic Cancer of the Colon or Rectum - International Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Principal Investigator, Dr. Naeem A. Chaudhri, Principal Investigator, King Faisal Specialist Hospital & Research Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAC #2041-082
Record Dates: First submitted 2007-10-01; First posted 2007-10-02 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-12

CONDITIONS: Colonic Neoplasms; Rectal Neoplasms
Keywords: Colon and Rectum Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Drug Therapy; Bevacizumab

INTERVENTIONS:
Radiation: First-Line Bevacizumab and Chemotherapy — Chemotherapy
Drug: Bevacizumab — Chemotherapy

SUMMARY:
First-Line Bevacizumab and Chemotherapy in Metastatic Cancer of the Colon or Rectum

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic cancer of colon or rectum

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Effectiveness | overall

SECONDARY OUTCOMES:
Quality of life | overall

CONTACTS AND LOCATIONS:
Overall Officials: Shouki Bazarbashi, MD, Principal Investigator — KFSH & RC